CLINICAL TRIAL: NCT06782230
Title: ScATtEred Rare Disease Biobanks: a Model of Sample/Data Collection With susTainablE and Shared Criteria SATELLITES
Brief Title: ScATtEred Rare Disease Biobanks: a Model of Sample/Data Collection With susTainablE and Shared Criteria
Acronym: SATELLITES
Status: Recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Sponsor
Other Study IDs: PNRR-MR1-2023-12377307; PNRR-MR1-2023-12377307 (Other Grant/Funding Number: Ministero della Salute)
Record Dates: First submitted 2024-10-11; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-09

CONDITIONS: Creation of an Italian Network of Biobanks of Rare Diseases
Keywords: Neuromuscolar disorders; Biobanking; Biological samples; Clinical data; Rare Diseases; Marfan Syndrome; Huntington disease; Angioedema; Congenital Heart Disease
MeSH Terms: conditions — Rare Diseases; Marfan Syndrome; Huntington Disease; Angioedema; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood samples will be collected and stored in biobanks to be used in future studies not yet defined.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rare diseases (RDs) have been defined by the European Union (EU) as life-threatening or chronically debilitating conditions affecting less than 1 person in 2000. RDs are complex and often need special treatments, thus combined efforts are required to address them to improve diagnosis, care and prevention. To date, over 6.000 RDs are known and most of them are "orphans". They do not have a market large enough to gather support to sustain research and discover treatments. Most RDs are disabling, incurable, painful and cause great suffering. Their complexity and heterogeneity often make diagnosis difficult; 25% of RD patients experience a diagnostic delay of 5 to 30 years and this has important implications for patient care. Thus, new diagnostic and therapeutic strategies are urgently needed. RDs registries are increasingly recognized as an effective tool to advance RD research. They are necessary to bring together patients and to pool data to achieve a sufficient sample size to facilitate epidemiological and/or clinical research. It is well known that registries are more effective when annexed to biobank infrastructure since make an important contribution to identify and validate biomarkers, uncover novel genes, elucidate pathogenesis at the Omics level, and develop new therapeutic strategies. Biobanks serve as biological samples and related clinical data repositories from affected patients and from undiagnosed patients experiencing with the "diagnostic odyssey", with the view of a retrospective diagnosis. The aim of creating a biobank is to make available a significant number of well-characterized and properly preserved samples and related data, to the scientific community for large-scale studies. Indeed, the recent advances in the technology of molecular biology and genetics require a large number of properly preserved biospecimens. This is certainly facilitated by building biobank networks. To this regard, in Italy, the collection of RDs samples is fragmented. The existing RD biobanks are of small or medium-size. They are stand-alone collections since only a limited networking among these infrastructures has been organized up to now. The objectives of this project will be: Aim 1: Establishment of the Scattered RD Biobank as a network of RD biobanks in order to overcome RD biological sample scarcity and to collect samples and data of high quality available to the scientific community for future collaborative studies in national and international co-operations Aim 2: Harmonization, Standardization and Network Governance. According to the document ISO 20387 illustrating the general requirements for biobanking, Standard Operating Procedures (SOPs) will be defined to ensure that every biobank in the network strictly follows the entire processes of collection, preparation, storage and distribution of biological material as well as related information and data. Common data bases and ethical/legal documents will be also generated. Aim 3: RD biobank upgrading and creation of novel RD biobanks. Already existing RD biobanks will be implemented in terms of organization of the sample collections according to the common SOPs and of extension of the sample collections and novel RD biobanks will be created such as Huntington's disease (OU3 and OU4), Marfan Syndrome, Hereditary Angioedema and Congenital Heart Diseases (OU1) biobanks. All the OU participating to this project are Reference Centre or Biological Research Centre (BRC) for RDs.

DETAILED DESCRIPTION:
Specific aim 1. Establishment of the Scattered RD Biobank. The aim of our project is to create the Scattered RD biobank as a network of novel dedicated and already existing biobank in order to overcome RD biological sample scarcity and to make high quality material available for future collaborative studies in national and international cooperation. The network will include mainly biobanks focused on cardiovascular and neurological RDs. It will be organized according to a bidirectional Hub&Spoke model in which each RD biobank serves as a centralised hub for samples and data collected from RD patients who refer to its own Institution/Centre and as a spoke for the other RD biobanks of the network. Each biobank will serves as hub for sample/data collection from RD patients who refer to other RD reference centres scattered throughout the territory and which do not have organized biobank according to the modern definition of biobank. This approach will favours the connection of different biobanks geographically spread through the Country and will avoid patient migration towards the biobank of interests. Two principal hubs will be defined: the Northern Hub to which the RD biobanks and RD Reference Centres of northern Italy will refer; and the Southern Hub to which the RD biobanks and RD Reference Centres of central and Southern Italy will refer. A Biospecimen Inventory Catalogue will be created and the description of all the procedures used for these collections (SOPs, sample associated data, ethical and legal documents) will be related to each sample and data.

Specific aim 2. Harmonization, Standardization and Network Governance. According to ISO 20387 that illustrates the general requirements for biobanking, Standard Operating Procedures (SOPs) will be defined to ensure consistency and standardization of practice (collection, preparation, storage and distribution of biological material as well as related information and data) in each single biobank. The biological samples from RD patients collected in the Scattered RD Biobank will be obtained following the specific SOPs generated for the collection of RD biological samples suitable for Omics approaches. SOPs will be generated for every stages of the pre-analytical process from collection to storage and more for the sharing of samples. The creation of the Scattered RD Biobank as biobank network needs of a rigorous Quality Management System (QMS) which is necessary to minimize inter-laboratory and intercentre variation and to guarantee the quality of the sample to be distributed in the collaborative projects. The QMS includes: (1) Quality Assurance to standardize all stages of the biobanking process, (2) Quality Controls (QC) on samples in order to validate the sample management process, to ensure reproducible quality and to the reliability of the storage procedures and the stability of the samples over time. QC will be performed both on the historical and new collections of RD biological samples to maximize experiment success and reliable interpretation of results. Sample QC will give valuable information to take preventive or corrective measures early, saving costs and reducing the risk of experimental errors. The most appropriate tools (markers and assays) that can be used to assess pre-analytical variations for both fluid and solid tissuederived samples will be defined for a better standardization between RD biobank laboratories. Data on biological samples and clinical information corresponding to the samples will be collected using a common database. The objective will be to harmonize and standardize the rules of communication between RD biobanks on the level of information about the donor and to facilitate sample location and access. To address these issues, a communication protocol according to MIABIS will be designed for the minimum information required to initiate collaborations among biobanks and to enable the exchange of biological samples. To facilitate harmonization of the different biobanks in the network, common regulations and fundamental ethical and legal documents will be also elaborated. Moreover, a website of the biobank network will be created to increase the visibility of the tool and to share all the elaborated documents. The website will include a "virtual biobank", an online catalogue of biological specimens stored in the biobanks. The virtual biobank will quickly and efficiently help investigators to find biospecimens that are located in different biobanks and will promote transparent sharing of bioresources in order to facilitate national and international collaborations. Specific aim 3.RD biobank upgrading and creation of novel RD biobanks. The already existing RD biobanks in the network will be implemented in terms of numerosity of samples collected and organization of the sample collections according to the common SOPs. All samples will be linked to relevant personal and health information, including health records, family history and lifestyle. They will be further characterized through genome data analysis and the phenotype regularly updated through follow-up visits. Novel biobanks will be established and dedicated to biological material and associated data deriving from subjects carrying Huntington disease (HD) mutations, Marfan Syndrome (MS), Hereditary Angioedema (HAE) and Congenital Heart Diseases (CHD). HD is a rare genetic neurodegenerative condition that today affects 1 out over 10,000 persons in Europe. The disease affects more than 6,000 people in Italy and around 40,000 people are considered 'at risk' of developing symptoms later in life. Although the disorder is well studied and characterized, much remains to be investigated on the diversity of symptoms among patients even within the same family. To this regard, the Centre for Rare Diseases of IRCCS Neuromed and the Untà Ricerca e Cura Huntington e Malattie Rare of IRCCS CSS are both recognized as reference centers for the disease at a national and international level. LIRH Foundation is a European HD Network site connected with HD family organizations across the Country. Its collaboration will guarantee the collection of clinical data which will be stratified according to disease stage and origin of samples from all over Italy. MS is a rare genetic condition happening in about 1 in 5,000 people and it is caused by a mutation in a gene called FBN1. MS affects connective tissue but it damages the blood vessels, heart, eyes, skin, lungs, and the bones of the hips, spine, feet and rib cage. Some complications of MS can be very serious, like an aneurysm (bulge) of the aorta. HAE is a rare, genetic disease characterized by unpredictable, recurrent episodes of skin and mucosal swelling most commonly caused by C1-inhibitor deficiency. The prevalence of HAE is estimated to be approximately 1 in 50,000 people worldwide. IRCCS Policlinico San Donato is a member of the ERN Guard Heart network, member of ITACA (Italian Network for Hereditary and Acquired Angioedema) and the headquarters of Cardio Vascular Genetics Centre. The establishment of a dedicated biobanks, will be an innovative and valuable tool for exploring genotype-phenotype correlations and molecular mechanisms underlying such a large variability. The establishment of these novel RD biobanks, will significantly impact on the national and international competitiveness of Italian biomedical research. The advantage of creating this kind of biobanks will result in having the possibility to collect multiple biological samples over the time during disease progression for each single subject. The function of the Scattered RD Biobank as research resource calls into question the processes and practices for recruitment, participation and engagement. The role of biobank participants is often passive after the initial enrolment and sample collection. However, to improve transparency and to demonstrate trustworthiness of the biobanks of the network, participants will be actively involved beyond the initial face-to-face towards more interactive dialogues with the research teams. Considering biobanking as a service for patients, a collaboration between RD biobanks of the network and Patient Organisations will be defined promoting dedicated meetings, round-tables and focus groups. A strong collaboration between RD biobanks and Patient Organisations will be also crucial to achieve the integration of sample data stored in biobanks and clinical data stored in registries or clinical databases.

WP1. Hub&Spoke model. The Scattered RD biobank will be created as a network of already existing and novel dedicated biobank mainly focused on cardiovascular and neurological RDs, according to a bidirectional Hub&Spoke model. The model will include two principal hubs, the Northern Hub and the Southern Hub , which already have experience in establishing of biobank networks. The objectives of these principal hubs will be: 1. To coordinate the creation of the Scattered RD biobank through the standardization and harmonization of all the procedures of the biobanking process.

Standard Operating Procedures (SOPs) for collection, processing and storage, quality control management, Ethical Legal Social Issue (ELSI) and uniformity in governance will be generated since biobanks will act as a single entity. 2. To manage and facilitate the connection of different biobanks and RD Reference Centres geographically spread through the Country. Virtual and in presence meetings between the representatives of the biobanks and of the RD Reference Centres will be periodically organized. 3. To be reference biobanks for RD Reference Centres scattered throughout the territory which do not have the facilities to collect samples and data for research studies, or for RD Reference Centres which have already collected samples and data but do not have a modern defined biobank and wish to be part of the Scattered RD biobank.

OU1 will be reference biobank of RD Reference Centres of Northern Italy and OU3 of RD Reference Centres of Central and Southern Italy. 4. To coordinate the creation of a Biospecimen Inventory Catalogue of samples/data collections already present in the biobanks of the network. A questionnaire will be generated and shared among the Units participating to this project and to the new biobanks or RD Reference Centres that desire to be part of the network. Questions will regard both information on the biobank infrastructures and facilities of the institution where the collection are stored and on the historical samples/data collections (SOPs developed and used for the collection, processing and storage, type of samples and associated data collected, number of patients involved, ethical and legal documents used, Quality Assurance policies). Moreover, the bidirectional model will plan that each Unit will be a centralised hub for historical and new collections from RD patients who refer to its own Institution/Centre and will be also a spoke for the network. Each Unit will collect and store new biological samples and associated data of patients with RDs and syndromes according to the SOPs and to the policies elaborated. Each Unit will be responsible of their own samples/data collection and will manage them according to the network governance.

WP2. Quality Manual: i) procedures for samples processing (e.g. aliquoting, storage and QC), supplies, equipment, instruments, reagents and labels; ii) procedures for obtaining informed consent and withdrawal of consent from participants; iii) management policies, including access control, backup systems, clinical annotation, document maintenance and archiving; iv) procedures for sample sharing and receiving, including methods and equipments; v) procedures for cost recovery; vi) organizational requirements (governance).

WP2.1 SOPs for the biobanking workflow according to official guidelines: 1. pre-analytical conditions (collection, initial processing, provisional cryopreservation of derivatives, long-term storage, testing) determined for each type of samples and derivatives; 2. selection of type of primary collection container (anticoagulant, preservative) and QRcoded cryotubes; 3. determination of the number and volume of sample aliquots; 4. procedures for distribution of samples using certified transportation companies.

WP2.2. Governance with the support of a Data Protection lawyer expert on legal biobank management: 1. sample access policy to provide researchers with a simple and transparent mechanism for accessing and sharing samples; 2. Steering Committee (PIs, biobank and RD Reference Centre managers, patient organization representative) will review all the requests for samples and related data and suggest approval, rejection or deferral; 3. Material Data Transfer Agreement (MDTA) to: i) govern the conditions under which the samples/data can be used; ii) outline the type of samples/data to be transferred, the purpose of the transfer, all restrictions or obligations related to the use of the samples and data; 4. ELSI issues to protect biobank donors and their personal data: i) creation of an Informed Consent according to the EU GDPR to offer to the donors sufficient information about benefits/risks of sample biobanking, to give them the possibility to revoke the consent, to assure them that their samples and data will be protected against misuse, will be safely stored and used for research. WP2.3. QMS: 1. QA guaranteed by the Quality Manual, by the definition of all non-conformities of primary samples or of derivate (e.g. haemolytic or lipemic blood, presence of clots) and by the traceability of sample and related information; 2. QC on samples to assess the quality of samples objectively and to validate the sample management process will be guarantee through: i) absolute assessment of the quality of samples; ii) suitability test. QC analyses on new and historical samples will be centralized in order ensure consistency in processes, share tools and best practices and impose some autonomy to the quality efforts as well as to provide strong quality system. WP3. Centralized database to improve the administration of samples collected in each biobank based on an integration between each biobank database software and the centralized database software. A minimum data set designed according to Minimum Information About Biobank data Sharing (MIABIS) will define: i) the biobank where the samples are stored; ii) the sample collection; iii) details on samples (e.g. sample type, storage temperature, anatomical site); iv) sample donor (e.g. date of birth, sex); v) event related to sample or donor (e.g. age at sampling, disease ontology, disease diagnosis). WP4. Website to increase the visibility of the biobanks and to share all the documents: i) public area accessible to all citizen that will contains general network information and contacts, news, events organized, study results; ii) catalogue of biological material stored to help investigators of other Institution to find samples of interest; iii) login reserved area accessible only to representative of each biobank of the network. Its creation will be performed by an agency specialized in web design and development of biobank websites.

WP5. Historical collections will be remodelled ad reorganized according to the activities described in this project in order to create the Biospecimen Inventory Catalogue designed to provide a list of all biospecimens and associated data already stored in the biobanks. Moreover, RD biobanks will implement the number of their samples and related data collecting new samples/data according to the Scattered RD Biobank SOPs generated and shared with the partners.

WP5.1. Based on the experience of already existing Italian RD biobank networks, the Scattered RD Biobank will promote the active participation of Patient Organizations in the establishment of this biobank network since it will represent a fundamental service for patients. Dedicated meetings and roundtables will be organized with the participation of biobankers, researchers, RD patient organization representatives, patients and relatives in order to discuss and share the biobank documents generated on policies and procedures, including those concerning ELSI issues. Moreover, meetings with experts of several biobanking aspects (healthcare professionals, bioethicists, DPO lawyers) will be organized to discuss on ethical and legal topics concerning privacy, informed consent, withdrawal of consent, samples and data access, return of results and incidental findings and where the patients and their relatives will have the opportunity to express their opinions, needs and expectations. Focus groups will be also organized with expert mediators to explore the opinions, knowledge, perceptions, and concerns of participants in regard to biobanking.

DATA COLLECTION AND MANAGEMENT. The minimum data set of standard attributes will define biobank and biological sample information (e.g. the biobank where the samples are stored, the sample collection, sample type, storage temperature, anatomical site) and donor information (e.g. date of birth, sex, age at sampling, disease ontology, disease diagnosis). All data will be recorded in the database software already present in the Units. In each RD Reference Center data collection will be conducted under the supervision of the Biobank Manager and of the PI that will have the responsibility to protect data security and privacy according to the institutional policies. All donors and related samples/data will be pseudonymized with an alphanumeric code. The minimum data set of each biobank will flow to a centralized database system based on an integration between each biobank database software and the centralized database software. This integration will be based on data exposure via API rest on TLS encrypted protocol. Due to the duration of the project, this integration will be implemented for the four Units participating to this project in order to build and test the architecture that could be extended to all biobanks in future projects. Regarding the previous collections, data will be re-organized according to the minimum data set generated.

BIOLOGICAL SAMPLES. New biological samples will be collected, processed, stored and shared according to the SOPs. Samples types collected will depend on the research projects (whole blood and derivates, FFPE or frozen tissues).

Samples will be divided in a defined volume and number of aliquots and stored in the biobanks partners. Regarding the historical collection, a Biospecimen Inventory Catalogue will be created and the description of all the procedures used for the collection (SOPs, sample associated data, ethical and legal documents) will be related to each sample and data.

SAMPLE QUALITY CONTROLS. 1. Absolute assessment of the quality of samples. Blood sample derivates: haemoglobin presence in plasma or serum, presence of cells or cell debris in plasma or serum, presence of platelet in plasma platelet free, cytofluorimetric analysis of the PBMC. Tissues: histological analysis of tissue stained slides to verify tissue architecture, cell morphology and sharpness. Nucleic acid samples: purity is calculated from the ratio of the absorbance measured by a spectrophotometer contributed by the nucleic acid to the absorbance of the contaminants. Typical requirements for A260/A280 ratios are 1.8¿2.2; A260/A280 of pure DNA is ~1.8, and A260/A280 of pure RNA is ~2.DNA/RNA integrity is evaluated by capillary electrophoresis techniques and represented by DNA/RNA Integrity Number DIN/RIN (where 1 indicates highly degraded DNA/RNA and 10 represents highly intact DNA/RNA). 2. Suitability test. Analysis of specific markers performed on the batch of the study samples to assess the fitness-for-purpose of samples, since a sample can be of high enough quality for one type of analysis (e.g., antibody analysis), but not for other types of analyses (e.g., metabolite analysis). QC of samples will be performed both on historical and new collection on randomly selected samples and if the quality did not meet the predefined criteria, corrective actions will be performed before continuing with the biobanking, in order to ensure a robust and reproducible process. For what concern the historical collections, the effect of freeze-thaw cycles and of different pre-storage handling conditions will be assessed and samples that fail to meet the quality control standards, will not be included. Intra-biobank QC samples will be performed to verify the QM of the single biobank samples assessing differences between separate studies on the same type of sample, and interbiobank QC samples will be performed to verify the QM of each biobank and to assess differences between the individual biobanks of the Scattered RD Biobank.

STATISTIC PLAN. In this project samples and data will be collected to be stored in the Scattered RD Biobank. No biological analyses will be performed on samples and no systematic examination, interpretation, and synthesis of collected clinical data will be performed to draw meaningful conclusions. A descriptive statistical analysis of data will be performerd in order to monitor the biobanking process. Descriptive statistical analysis will be expressed in terms of mean (standard deviation) or median (range, interquartile range) for continuous variables and as absolute and relative frequencies for categorical variables Comparisons between two independent groups will be made by unpaired T-test or Wilcoxon sum rank test as appropriate.

Inferential procedures (hypothesis testing and confidence intervals) and regression models will also be properly applied depending on the purpose of each specific analysis. Quality Control. A sample size of 325 from a batch of 2000 allows to evaluate 5% of risk of rejecting sample and 5% of risk of accepting a sample nonconforming, based on an acceptable quality level of 5% and a limiting quality level of 2%. The acceptance cutoff number is 8.

EXPECTED OUTCOMES. 1. Establishment of the Scattered RD Biobank through i) harmonization and standardization of the biobanking process of the biobanks of the network; ii) the realization of the Quality Manual of the Scatterd RD Biobank containing SOPs for collection, preparation, storage and distribution of the biological material/data, common regulations and fundamental ethical and legal documents (e.g. informed consent, MDTA) and the Quality Management System; iii) the creation of a centralized database with a minimum data set. 2. Development of Quality Control (QC) systems on biological samples in order to ensure the creation of high-quality collections. QC systems include specific tests and analyses to be performed on biological samples and the definition of cutoff values for acceptance in Scattered RD Biobank of historical or new collections. 3. Creation of Biospecimen Inventory Catalogue of samples/data collected by the single biobanks before the establishment of the network that allows a better management and valorisation of historical collections. This leads to an increase the utilisation rates of the samples/data collected and reduce the volumes of specimens stored. The biobanks of the network will be more selective as to what they stored assisting to a transition from a biobanking model based on mostly retrospective samples of pre-defined specimens to a more prospective, investigator-driven collection in order to reduce cost of duplicate collections. 4. Increase the visibility of biobanks creating a website of the network to improve the sharing of sample/data collected and to facilitate the access of biobanks and RD Reference Centers to national and international research projects. On the website, potential stakeholders can find the ¿virtual biobank¿ of the Scattered RD Biobank with the catalogue of the biological specimens of the network.

5. Establishment of the collaboration between Patient Organizations and the Scattered RD Biobank thanks to formal agreement. The effective collaboration between patients and the scientific community is essential to the enhancement of awareness and trust, as well as to the sharing of objectives and efforts to support research on RD 6. Identify and include in the Scattered RD Biobank singles and small biobanks that are not yet part of any network and are stand-alone collections without a policy for cross-border sharing of samples or specific workflows implemented to guarantee the quality of the biological sample and of the associated data collected. Be part of Scattered RD Biobank will help these biobanks to evolve from a biobank focused on the number of samples collected to a biobank focused on the quality of biospecimens and data.

RISK ANALYSES. This two-years research grant will cover the costs of the establishment of the Scatterd RD Biobank and of the start-up of infrastructures. However, the Scattered RD Biobank is a long- term project that needs longitudinal economic sustainability. The biobanks partners of this network are located within scientific institutions, that will guarantee financial cover of basic activities, such as the m aintenance of equipment servicing and utility bills, e.g. for electricity and gases, which are largely consumed by the freezing systems. However, the economic sustainability of the Scatterd RD Biobank might a bottleneck due to the maintenance costs. Managerial solutions for the long-term sustainability of the network should be: i) to access to national and international funding mechanisms for RD project grants; ii) to introduce cost recovery procedures for sample acquisition, storage, and handling. Indeed, costs of biospecimen acquisition, procuring, processing storage, and preserving represent a substantial proportion of the total expenses by a biobank; (iii) to increase the number of samples distributed.

The rate of samples storing should not grow faster than utilisation rates; iv) to engage with multiple types of stakeholders, such as patient associations and donors, hospitals and clinicians, researchers, public administration and charities; v) to improve understanding of the biobank benefits for the economy and society since biobanks play a central role in improving patient diagnosis and therapeutic care and thus enhancing public and private fundings.

The development of Scattered RD Biobank is not trivial due to heterogeneity of the biobanks/RD Reference Centers in samples and data collection. Harmonized guidelines should be generated to organize historical and new sample/data collections in terms of biobanking procedures, data protection, sample/data sharing and databases. Database softwares, such as biobank information management systems (BIMS), harmonized services and common ontologies (MIABIS) should be used to allow interoperability of data and sample collections. The quality of biobanks depends significantly on the work of the adequately trained personnel, who is responsible for the reception, processing and storage of biosamples and related data. The biobank personnel must guarantee a consistent sample quality fundamental for the success of the single biobank and thus of the network. Recruiting personnel for a project of this dimension is crucial to reach the full potential, especially for biobanks needing new personnel¿s recruitments. Harmonised training for technical staff should be provided for the success of the network project since neglecting employees¿ training measures can damage public health and should be a risk of damaging the reputation of the biobanks and host institution. New staff will be appropriately trained before becoming fully integrated into the work environment learning about teamwork, personnel safety, patient privacy, samples quality, and best practices in the form of carefully implemented SOPs.

Harmonization has a key role in the establishment of a biobank network but many ethical and legal problems have to be resolved. Expert on ethical and legal frameworks and national legislation will be invited to participate in the whole process of development of biobank networks, to provide protection of donors and ensure appropriate use of their samples.

ELIGIBILITY:
Inclusion Criteria: patients with a rare disease or family members -

Exclusion Criteria: none

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The biobank network will collect samples from subjects affected by rare diseases mainly Huntington disease (HD), Marfan Syndrome (MS), Hereditary Angioedema (HAE) and Congenital Heart Diseases (CHD). Samples from other type of rare diseseas will be also collected
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-08-31 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Establishment of the Scattered RD Biobank | 24 months
  Establishment of the Scattered RD Biobank

CONTACTS AND LOCATIONS:
Overall Officials: Rosanna Cardani, PhD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- BioCor Biobank IRCCS-Policlinico San Donato, San Donato Milanese, Milan, Italy